CLINICAL TRIAL: NCT05934201
Title: Futbolcularda Bel Ağrısının ve Motor Kontrol Etkileniminin Sportif Performansa Etkilerinin İncelenmesi
Brief Title: Low Back Pain and Motor Control in Soccer Players
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Associate Professor, Hacettepe University
Other Study IDs: GO 22/110
Record Dates: First submitted 2023-04-05; First posted 2023-07-06 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low-back Pain
Keywords: soccer; motor control; balance; agility; performance; coordination; speed; functional movement screen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identification of the effects of low back pain and motor control influence on soccer players performance.

DETAILED DESCRIPTION:
At least 60 volunteer athletes who playing soccer at least 3 years, not away from field more than 2 weeks, 16 years and older are planned to include this study. All participating athletes in this study will be signed an informed consent form then their demographic information will be recorded. To evaluate disability due to low back pain, musculoskeletal problems and the willingness to participate in sports will be used the Oswestry Disability index, the Nordic Musculoskeletal System questionnaire and the Sport Motivation Scale-2, respectively. The motor control levels of the athletes will be assessed with the motor control test battery (MKTB), the core stability with the Sahrmann's core stability test, core muscles endurance with the sport-specific endurance plank test and side bridge endurance test, the static balance with the stand stork test, the dynamic balance with the lower quadrant y balance test, postural changes with the Corbin Posture Rating Scale, the agility with the T test, speed and coordination with 4-10 shuttle run test, explosive force with long jump test, the kinetic chain with the functional movement screen.

ELIGIBILITY:
Inclusion Criteria:

* Be over 16 years old,
* Participating in the soccer training for at least three years,
* Soccer players who have not stayed away from their sport for more than two weeks

Exclusion Criteria:

* Any history of orthopedic or neurological injury or pain that may interfere with normal football training or competition during assessment
* History of spine/lower and upper extremity surgery,
* Structural deformities such as scoliosis and kyphosis,
* Having trap neuropathy
* Soccer players who had injuries other than chronic low back pain in the last 6 months will be excluded from the study.

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: All volunteer employees who are over the age of 16, have been playing football for at least three years, have not been away from football for more than two weeks, play football and meet the inclusion criteria of the study will be included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor control disorder | baseline
  Motor control test battery: the test consists of ten different tests (forward bend, return from forward bend, sitting forward lean,sitting knee extension, pelvic tilt, one leg stance,side bending, rocking forward, prone knee flexion, hip abduction).Whether the total score increases, the motor control disorders increase.
Core stability | baseline
  Sharmann's core stability test
Core muscles endurance | baseline
  Sport-specific endurance plank test, right and left side bridge endurance test
Static balance | baseline
  Stand Stork test
Dynamic balance | baseline
  Lower quadrant y balance test
Agility | baseline
  T test
Speed and coordination | baseline
  4-10 Shuttle run test
Explosive power | baseline
  Standing long jump test
Kinetic chain | baseline
  Functional movement screen

SECONDARY OUTCOMES:
Nordic Musculoskeletal System Questionnaire | baseline
  Evaluates the musculoskeletal system problem. If the athlete indicate a musculoskeletal problem different than low back pain, it will use for screening.
Sport Motivation Scale-2 | baseline
  Evaluates willingness to participate in sports. The scale has 6 subparameters indicating sport motivation levels is high or low.
Oswestry Disability Index | baseline
  Evaluate disability due to low back pain. the index measures perceived low back pain related dysfunction. Whether the total score increaeses, the dyscfunction increases.
Postural changes | baseline
  Corbin Posture Rating Scale. Whether the total score increaeses, thepostural problems increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Aynur Demirel, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Akkus C, Demirel A. The impact of chronic low back pain and motor control impairment on athletic performance in elite soccer players: a cross-sectional study. BMC Musculoskelet Disord. 2025 Aug 12;26(1):781. doi: 10.1186/s12891-025-09023-x. PMID 40797311